CLINICAL TRIAL: NCT01535326
Title: Comparing Air Insufflation, Water Immersion and Water Exchange Methods During Minimal Sedated Colonoscopy, a Randomized, Controlled Trial
Brief Title: Comparing Water Immersion and Water Exchange Methods During Minimally Sedated Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsi hsieh, Chief of department of gastroenterology and hepatology, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DalinTCGH-hsieh-01
Record Dates: First submitted 2012-02-11; First posted 2012-02-17 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Colon Neoplasm; Pain
Keywords: colonoscopy
MeSH Terms: conditions — Colonic Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- air insufflation (Placebo Comparator): Use air insufflation during colonoscopy
  Interventions: Procedure: air insufflation
- water immersion (Active Comparator): infuse water during insertion, remove water during withdrawal of colonoscopy
  Interventions: Procedure: water immersion
- water exchange (Active Comparator): infuse and remove water during insertion phase of colonoscopy
  Interventions: Procedure: water exchange

INTERVENTIONS:
Procedure: air insufflation — insufflate air during the insertion of colonoscopy
  Arms: air insufflation
Procedure: water immersion — infuse water during insertion, aspirate water during withdrawal
  Arms: water immersion
Procedure: water exchange — infuse and remove water during insertion phase of colonoscopy
  Arms: water exchange

SUMMARY:
In minimally sedated Asian patients in a community setting the investigators showed that a limited volume of water infusion instead of air insufflation in either the rectal sigmoid colon or the whole colon significantly reduced pain score during colonoscopy. Cecal intubation rate was not compromised. The reduction of pain score ranges from 25% to 32 % in our previous studies.1, 2 In contrast, several US reports described the successful use larger volumes of water infused throughout the entire colon in patients undergoing colonoscopy which result in a greater reduction of the pain score, averaging about 56%.3-5 A recent review suggested that the cause of the difference might lies in the timing of water removal.6 Specifically, the investigators group removed the infused water predominantly during withdrawal phase (water immersion) and the U.S. group removed water during insertion phase (water exchange).

This prospective, randomized controlled trial compared water exchange or water immersion with traditional air insufflation in patients undergoing minimally sedated colonoscopy. The investigators test the hypothesis that water exchange can reduce more pain than water immersion in the investigators clinical setting.

DETAILED DESCRIPTION:
All procedures will be recorded and stored as digital files.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing minimally sedated colonoscopy

Exclusion Criteria:

* Obstructive lesions of the colon, inadequate bowel preparation, allergy to meperidine, massive ascites, past history of partial colectomy, or refusal to provide written informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, Dr., Principal Investigator — Dalin Tzu Chi General Hospital
Locations (1):
- Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Hsieh YH, Lin HJ, Tseng KC. Limited water infusion decreases pain during minimally sedated colonoscopy. World J Gastroenterol. 2011 May 7;17(17):2236-40. doi: 10.3748/wjg.v17.i17.2236. PMID 21633535
- [Background] Leung F, Harker J, Leung J, Siao-Salera R, Mann S, Ramirez F, Friedland S, Amato A, Radaelli F, Paggi S, Terruzzi V, Hsieh Y. Removal of infused water predominantly during insertion (water exchange) is consistently associated with a greater reduction of pain score - review of randomized controlled trials (RCTs) of water method colonoscopy. J Interv Gastroenterol. 2011 Jul;1(3):114-120. doi: 10.4161/jig.1.3.18510. Epub 2011 Jul 1. PMID 22163081
- [Background] Leung J, Mann S, Siao-Salera R, Ransibrahmanakul K, Lim B, Canete W, Samson L, Gutierrez R, Leung FW. A randomized, controlled trial to confirm the beneficial effects of the water method on U.S. veterans undergoing colonoscopy with the option of on-demand sedation. Gastrointest Endosc. 2011 Jan;73(1):103-10. doi: 10.1016/j.gie.2010.09.020. PMID 21184876
- [Background] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Air Insufflation | Water Immersion | Water Exchange
Started | 90 | 90 | 90
Completed | 90 | 90 | 90
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients underwent endoscopy by YHH
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Insufflation | Water Immersion | Water Exchange | Total
Number analyzed (Participants) | 90 | 90 | 90 | 270
Age, Continuous [Median (Full Range); unit: years] | 59 [25 to 78] | 53 [28 to 79] | 58 [23 to 77] | 55 [23 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 35 | 102
  Male | 60 | 53 | 55 | 168

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Without Pain
Description: proportion of patients without insertion pain during colonoscopy
Time Frame: up to 12 months
Measure: Number; unit: participants
Groups:
- Air Insufflation: Use air insufflation during colonoscopy
  air insufflation: insufflate air during the insertion of colonoscopy
  Proportion of no pain: 30%
- Water Immersion: infuse water during insertion, remove water during withdrawal of colonoscopy
  water immersion: infuse water during insertion, aspirate water during withdrawal
  Proportion of no pain: 43.3%
- Water Exchange: infuse and remove water during insertion phase of colonoscopy
  water exchange: infuse and remove water during insertion phase of colonoscopy
  Proportion of no pain: 61.1%
Arm/Group | Air Insufflation | Water Immersion | Water Exchange
Number analyzed (Participants) | 90 | 90 | 90
participants | 27 | 39 | 55

2. Secondary Outcome: Patient Pain Score
Description: The maximal pain score during insertion phase of colonoscopy was assessed with 0 to 10 scale VAS score (0: no pain; 10: maximal pain)
Time Frame: 9 to 12 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Air Insufflation | Water Immersion | Water Exchange
Number analyzed (Participants) | 90 | 90 | 90
units on a scale | 3.5 [0 to 10] | 1.8 [0 to 8.5] | 0 [0 to 10]

3. Secondary Outcome: Patient Satisfaction Score
Description: satisfaction score obtained after colonoscopy 0 = no satisfied; 10 = most satisfied
Time Frame: 9 to 12 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Air Insufflation | Water Immersion | Water Exchange
Number analyzed (Participants) | 90 | 90 | 90
units on a scale | 10 [6.5 to 10] | 10 [7 to 10] | 10 [8 to 10]

4. Secondary Outcome: Number of Participants With at Least One Adenoma
Description: the number of participants with at least one adenoma in each of the study groups.
Time Frame: 9 to 12 months
Measure: Number; unit: participants
Arm/Group | Air Insufflation | Water Immersion | Water Exchange
Number analyzed (Participants) | 90 | 90 | 90
participants | 39 | 41 | 51

5. Other Pre Specified Outcome: Post-procedure Discomforts and 30 Day Complication Rate
Description: telephone follow up for post-procedure discomforts and 30 day complication rate
Time Frame: one month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Air Insufflation | Water Immersion | Water Exchange
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 1/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Air Insufflation (N=90) | Water Immersion (N=90) | Water Exchange (N=90)
perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — one patient received polypectomy during withdrawal phase. Perforation was found immediately and hemoclips were applied. She recovered uneventfully after supportive care.

LIMITATIONS AND CAVEATS:
Single center; single endoscopist

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes